CLINICAL TRIAL: NCT03990649
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of TAK-935 as an Adjunctive Therapy in Adult Subjects With Chronic Complex Regional Pain Syndrome
Brief Title: Study of TAK-935 as an Adjunctive Therapy in Adult Participants With Complex Regional Pain Syndrome (CRPS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-935-2008
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Results first posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Complex Regional Pain Syndrome
Keywords: Drug Therapy; Soticlestat; TAk-935
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — soticlestat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Double-Blind Treatment Period - Part A: Placebo (Placebo Comparator): Soticlestat matching placebo tablets, orally, twice daily (BID) for Weeks 1, 2 and 3 in Double blind Titration Period. Soticlestat matching placebo tablets, orally BID for 12 weeks in Double blind Maintenance Period. Taper period (if participant did not continue to Part B): Dose of soticlestat matching placebo tablets was reduced to next lower dose every 3 days (maximum 6 days) until discontinuation.
  Interventions: Drug: Placebo
- Double-Blind Treatment Period - Part A: Soticlestat (Experimental): Soticlestat, tablet, orally, 100 mg BID for Week 1, followed by 2×100 mg tablets, soticlestat, orally BID for Week 2, further followed by 3×100 mg tablets, soticlestat, orally BID for Week 3. Dose was uptitrated every week based on safety and tolerability. Part A (Double blind Maintenance Period): 3×100 mg tablets, soticlestat, orally BID for 12 weeks. Dose was adjusted during Maintenance Period due to safety and tolerability. Taper Period (if participant did not continue to Part B): Dose of soticlestat was reduced to next lower dose every 3 days (maximum 6 days) until soticlestat was discontinued.
  Interventions: Drug: Soticlestat
- Open-Label Extension Period - Part B: Soticlestat (Experimental): Soticlestat, 2×100 mg tablets, orally, BID for Week 1, followed by 3×100 mg tablets, soticlestat, orally, BID for Week 2. Dose was uptitrated every week based on safety and tolerability. Part B (Open label extension: Maintenance Period): 3×100 mg tablets, soticlestat, orally, BID for 12 weeks. Dose was adjusted during Maintenance Period due to safety and tolerability. Taper Period: Dose of soticlestat was reduced to next lower dose every 3 days (maximum 6 days) until soticlestat was discontinued.
  Interventions: Drug: Soticlestat

INTERVENTIONS:
Drug: Soticlestat — Soticlestat tablets
  Other Names: TAK-935
  Arms: Double-Blind Treatment Period - Part A: Soticlestat; Open-Label Extension Period - Part B: Soticlestat
Drug: Placebo — Soticlestat matching placebo tablets
  Arms: Double-Blind Treatment Period - Part A: Placebo

SUMMARY:
The purpose of this study is to investigate the effect of soticlestat (TAK-935) on calculated 24-hour average pain intensity by the numeric pain scale (NPS).

DETAILED DESCRIPTION:
The drug being tested in this study is called soticlestat (TAK-935). Soticlestat is being tested to treat people with chronic complex regional pain syndrome (CRPS). This study will look at the efficacy, safety, and tolerability of soticlestat as an adjunctive therapy in participants with CRPS.

The study will enroll approximately 24 patients. Participants will be randomly assigned (by chance, like flipping a coin) in 2:1 ratio to one of the two treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

Soticlestat 100 mg tablets, 100, 200 or 300 mg twice daily (BID) Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient

Participants will receive 100 mg soticlestat tablets or soticlestat matching placebo tablets, BID for Week 1, 2x100 mg soticlestat tablets or soticlestat matching placebo tablets, BID for Week 2 and followed by 3x100 mg soticlestat tablets or soticlestat matching placebo tablets, BID for Week 3. Dose will be uptitrated based on safety and tolerability in titration period. Participants will continue to receive the same dose in maintenance period. Dose adjustments during maintenance period may take place due to safety and tolerability.

Participants will then enter Part B (optional) or taper period. In Part B all participants will receive soticlestat 2x100 mg tablets, BID for 1 Week, followed by soticlestat 3x100 mg tablets, BID for 1 Week. Dose will be uptitrated/downtitrated based on safety and tolerability in titration period (Part B), participants will continue to receive the same dose in maintenance period (Part B) and followed by a taper period.

This multi-center trial will be conducted in United Kingdom. The overall time to participate in this study is approximately 36 weeks. Participants will make multiple visits to the clinic and will be contacted by telephone 15 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Participant meets the Budapest clinical diagnosis of complex regional pain syndrome (CRPS) at the screening visit and is at least 6 months since onset of symptoms.
2. Participant's pain medications and nondrug treatments must be stable (regimented per prescription) for 1 month prior to screening and remain stable throughout Part A.
3. Participant agrees to use a single previously prescribed rescue medication within the prescribed dose during Part A of the study and to record the daily use of these medications.
4. Participant must have an average 24-hour pain intensity score ≥4 and ≤9 on the 24-hour average pain intensity numeric pain scale (NPS) during screening/baseline. This score will be calculated by averaging the daily 24 hour pain intensity scores for the past seven days prior to randomization. The participant must have daily 24-hour pain intensity scores recorded for at least 6 of the past 7 days.

Exclusion Criteria:

1. Currently receiving intravenous (IV) or oral ketamine, history of IV or oral ketamine use within the past 6 weeks prior to screening, or planned use of IV or oral ketamine during this study.
2. Participant is receiving chronic opioid treatment at a dose that has not been stable 28 days prior to screening.
3. Participant is receiving chronic opioid treatment >160 mg of morphine equivalent per day.
4. Participant has a positive drug screen for phencyclidine, amphetamine/ methamphetamine, or cocaine at screening. Cannabis is allowed..
5. Participant is positive for hepatitis B or hepatitis C infection at screening. (Note that participants who have been vaccinated against hepatitis B [hepatitis B surface antibody {Ab}-positive] who are negative for other markers of prior hepatitis B infection [eg, negative for hepatitis B core Ab] are eligible. Also, note that participants who are positive for hepatitis C Ab are eligible if they have a negative hepatitis C viral load by quantitative polymerase chain reaction).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- United Kingdom (3):
  - St Pancras Clinical Research, London, England
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston, England
  - University Hospital Southampton NHS Foundation Trust, Southampton, England

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Ratcliffe S, Arkilo D, Asgharnejad M, Bhattacharya S, Harden RN. Randomized controlled study to evaluate the efficacy and safety of soticlestat as adjunctive therapy in adults with complex regional pain syndrome. Pain Med. 2023 Jul 5;24(7):872-880. doi: 10.1093/pm/pnac198. PMID 36538782

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at three investigative sites in United Kingdom (UK) from 23 July 2019 to 28 October 2020.
Pre-assignment Details: Participants with a diagnosis of chronic complex regional pain syndrome (CRPS) were enrolled to receive soticlestat or placebo in Part A (Double-blind [DB] Treatment Period) and soticlestat in Part B (Open-label [OL] Treatment Period). Following completion of the Part A, participants had an option to continue into Part B.
Period: Part A: DB Treatment Period (15 Weeks)
Arm/Group | Double-Blind Treatment Period - Part A: Placebo | Double-Blind Treatment Period - Part A: Soticlestat | Open-Label Extension Period - Part B: Soticlestat
Started | 9 | 15 | 0
Completed | 6 | 12 | 0
Not Completed | 3 | 3 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Reason not Specified | 1 | 1 | 0
Period: Part B: OL Extension Period (14 Weeks)
Arm/Group | Double-Blind Treatment Period - Part A: Placebo | Double-Blind Treatment Period - Part A: Soticlestat | Open-Label Extension Period - Part B: Soticlestat
Started | 0 | 0 | 18
Completed | 0 | 0 | 14
Not Completed | 0 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Reason not Specified | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set for Part A included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind Treatment Period - Part A: Placebo | Double-Blind Treatment Period - Part A: Soticlestat | Total
Number analyzed (Participants) | 9 | 15 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (13.51) | 42.1 (10.27) | 41.0 (11.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 14 | 21
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 15 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 9 | 15 | 24
Numeric Pain Scale (NPS) Score [Mean (Full Range); unit: scores on a scale] — The 24-hour average pain intensity was calculated from current pain intensity scores collected three times a day as measured by the electronic pain diary daily using NPS. NPS is an 11-point scale, where scores range from 0-10, 0= no pain to 10 = most pain imaginable.
  scores on a scale | 6.33 [4.9 to 7.8] | 6.33 [4.5 to 7.6] | 6.33 [4.5 to 7.8]
Patient-Reported Outcomes Measurement Information System (PROMIS-29) Version 2.1 Domain Score [Mean (Standard Deviation); unit: t-score] — PROMIS-29 (v2.1) assess health-related quality of life for 7 domains with T-scores of reference population: Depression:1=never-5=always;T-scores:41.0-79.4. Physical function:1=unable to do-5=without any difficulty;T-scores:22.5-57.0 3. Anxiety:1=never-5=always;T-scores:40.3-81.6. Pain interference: 1=not at all-5=very much;T-scores:41.6-75.6.Fatigue:1=not at all-5=very much;T-scores:33.7-75.8. Sleep disturbance:1=very much-5=not at all;T-scores:32.0-73.3. Ability to participate in social roles and activities:1=always-5=never;T-scores:27.5-64.2 Higher scores=more of domain being measured.
  t-score
    Physical Function | 35.83 (5.607) | 34.65 (4.743) | 35.09 (4.998)
    Anxiety | 46.30 (11.906) | 51.94 (8.873) | 49.83 (10.248)
    Depression | 47.31 (12.523) | 47.27 (8.868) | 47.28 (10.120)
    Fatigue | 57.17 (8.427) | 60.55 (8.280) | 59.28 (8.321)
    Sleep Disturbance | 54.63 (3.854) | 54.99 (2.390) | 54.86 (2.945)
    Ability to Participate in Social Roles and Activities | 40.03 (6.205) | 39.11 (4.723) | 39.45 (5.213)
    Pain Interference | 66.37 (6.710) | 64.22 (8.039) | 65.03 (7.492)
CRPS Severity Score (CSS) Total Score [Mean (Standard Deviation); unit: scores on a scale] — Signs and symptoms reflecting the sensory, vasomotor, sudomotor/edema, and motor/trophic disturbances of CRPS had been incorporated into a clinically feasible CSS. Total CSS is a 16-point score which was calculated by the number of "yes" answers to the questions on the 8 symptoms and 8 signs when all 16 questions were answered.
  scores on a scale | 12.7 (1.73) | 12.9 (1.87) | 12.8 (1.79)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean 24-Hour Pain Intensity as Assessed by NPS Score to the End of Part A
Description: The 24-hour average pain intensity was calculated from current pain intensity scores collected three times a day as measured by the electronic pain diary daily using NPS. NPS is an 11-point scale, where scores range from 0-10, 0= no pain to 10 = most pain imaginable. Negative change from Baseline indicated improvement.
Time Frame: Baseline and Week 15
Population: Full Analysis Set for included all participants who were randomized, received at least 1 dose of study drug, and had at least one valid post-baseline value for the assessment of average 24-hour pain score. The data is reported for Part A in this outcome measure. Overall number of participants analyzed are the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Double-Blind Treatment Period - Part A: Placebo | Double-Blind Treatment Period - Part A: Soticlestat
Number analyzed (Participants) | 7 | 12
scores on scale | -0.74 (1.614) | -1.05 (1.310)

2. Secondary Outcome: Percent Change From Baseline in Mean 24-Hour Pain Intensity as Assessed by NPS Score to the End of Part A
Description: The 24-hour average pain intensity was calculated from current pain intensity scores collected three times a day as measured by the electronic pain diary daily using NPS. NPS is an 11-point scale, where scores range from 0-10, 0= no pain to 10 = most pain imaginable. Negative percent change from Baseline indicated improvement.
Time Frame: Baseline and Week 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Double-Blind Treatment Period - Part A: Placebo | Double-Blind Treatment Period - Part A: Soticlestat
Number analyzed (Participants) | 7 | 12
percent change | -12.20 (29.108) | -18.35 (23.699)

3. Secondary Outcome: Percentage of Participants Considered Responders at the End of Part A
Description: Response was defined as ≥ 30% improvement on the 24-hour pain intensity as assessed by the NPS score. The 24-hour average pain intensity was calculated from current pain intensity scores collected three times a day as measured by the electronic pain diary daily using NPS during Part A. NPS is an 11-point scale, where scores range from 0-10, 0= no pain to 10 = most pain imaginable.
Time Frame: Week 15
Population: Full Analysis Set for included all participants who were randomized, received at least 1 dose of study drug, and had at least one valid post-baseline value for the assessment of average 24-hour pain score. The data is reported for Part A in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Treatment Period - Part A: Placebo | Double-Blind Treatment Period - Part A: Soticlestat
Number analyzed (Participants) | 9 | 15
percentage of participants | 22.2 | 26.7

4. Secondary Outcome: Change From Baseline in Domain Score of PROMIS-29 Version 2.1 at the End of Part A
Description: PROMIS-29 (v2.1) is a health-related quality of life survey assessing 7 domains with 4 questions on a 5-point Likert scale. Total raw domain scores are converted into T-scores from a reference population: Depression: 1=never to 5=always, T-scores:41.0-79.4; Physical function: 1=unable to do to 5=without any difficulty, T-scores: 22.5-57.0; Anxiety: 1=never to 5=always, T-scores: 40.3-81.6; Pain interference: 1=not at all to 5=very much, T-scores: 41.6-75.6; Fatigue: 1=not at all to 5=very much, T-scores: 33.7-75.8; Sleep disturbance: 1=very much to 5=not at all, T-scores: 32.0-73.3; Ability to participate in social roles or activities: 1=always to 5=never, T-scores: 27.5-64.2. High scores signify more of domain being measured. Thus, on symptom-oriented domains, higher scores=worse symptomatology and a negative change from Baseline indicates improvement. On function-oriented domains, higher score=better functioning and a positive change from Baseline indicates improvement.
Time Frame: Baseline and Week 15
Population: Full Analysis Set for included all participants who were randomized, received at least 1 dose of study drug, and had at least one valid post-baseline value for the assessment of average 24-hour pain score. The data is reported for Part A in this outcome measure. Number analyzed are the number of participants with data available for analyses in the given category (domain).
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Double-Blind Treatment Period - Part A: Placebo | Double-Blind Treatment Period - Part A: Soticlestat
Number analyzed (Participants) | 9 | 15
t-score
  Physical Function: number analyzed (Participants) | 8 | 12
  Physical Function | 1.53 (2.207) | 2.39 (4.042)
  Anxiety: number analyzed (Participants) | 8 | 13
  Anxiety | 3.29 (10.348) | -1.99 (9.567)
  Depression: number analyzed (Participants) | 8 | 13
  Depression | 1.15 (10.011) | -0.78 (6.902)
  Fatigue: number analyzed (Participants) | 8 | 13
  Fatigue | 0.45 (12.126) | -3.66 (10.456)
  Sleep Disturbance: number analyzed (Participants) | 8 | 13
  Sleep Disturbance | 2.13 (5.110) | 2.55 (1.927)
  Ability to Participate in Social Roles: number analyzed (Participants) | 7 | 13
  Ability to Participate in Social Roles | 1.66 (6.051) | 2.74 (5.147)
  Pain Interference: number analyzed (Participants) | 7 | 13
  Pain Interference | -1.53 (6.257) | -0.38 (7.597)

5. Secondary Outcome: Percent Change From Baseline in Domain Score of PROMIS-29 Version 2.1 at the End of Part A
Description: as for outcome 4
Time Frame: Baseline and Week 15
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Double-Blind Treatment Period - Part A: Placebo | Double-Blind Treatment Period - Part A: Soticlestat
Number analyzed (Participants) | 9 | 15
percent change
  Physical Function: number analyzed (Participants) | 8 | 12
  Physical Function | 4.27 (6.197) | 8.00 (14.106)
  Anxiety: number analyzed (Participants) | 8 | 13
  Anxiety | 9.35 (24.153) | -2.43 (16.584)
  Depression: number analyzed (Participants) | 8 | 13
  Depression | 4.51 (21.864) | 0.04 (13.494)
  Fatigue: number analyzed (Participants) | 8 | 13
  Fatigue | 2.42 (22.902) | -4.62 (16.045)
  Sleep Disturbance: number analyzed (Participants) | 8 | 13
  Sleep Disturbance | 4.46 (9.611) | 4.75 (3.600)
  Ability to Participate in Social Roles: number analyzed (Participants) | 7 | 13
  Ability to Participate in Social Roles | 4.39 (15.195) | 7.42 (13.796)
  Pain Interference: number analyzed (Participants) | 7 | 13
  Pain Interference | -1.88 (9.149) | 0.82 (15.571)

6. Secondary Outcome: Percentage of Participants in Each Category of the Patient Global Impression of Change (PGIC) Scale at the End of Part A
Description: The PGIC is a 7-point Likert scale to address the following question: Since beginning treatment at this clinic would you describe any changes (if any) in activity, limitations, symptoms, emotions and overall quality of life related to your painful condition compared to before treatment? Participants select from scale range of 1-7: very much improved (1); much improved (2); minimally improved (3); no change (4); minimally worse (5); much worse (6); very much worse (7). Only categories with at least 1 participant were reported.
Time Frame: Week 15
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Treatment Period - Part A: Placebo | Double-Blind Treatment Period - Part A: Soticlestat
Number analyzed (Participants) | 9 | 15
percentage of participants
  Much Improved | 33.3 | 33.3
  Minimally Improved | 11.1 | 13.3
  No Change | 22.2 | 33.3
  Minimally Worse | 11.1 | 0
  Missing | 22.2 | 20.0

7. Secondary Outcome: Change From Baseline in Complex Regional Pain Syndrome (CSS) at the End of Part A
Description: Signs and symptoms reflecting the sensory, vasomotor, sudomotor/edema, and motor/trophic disturbances of CRPS had been incorporated into a clinically feasible CSS. Total CSS is a 16-point score which was calculated by the number of "yes" answers to the questions on the 8 symptoms and 8 signs when all 16 questions were answered. Negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Double-Blind Treatment Period - Part A: Placebo | Double-Blind Treatment Period - Part A: Soticlestat
Number analyzed (Participants) | 6 | 13
scores on scale | -2.2 (2.48) | -3.1 (3.12)
Statistical Analysis 1: Comparison: Double-Blind Treatment Period - Part A: Placebo vs Double-Blind Treatment Period - Part A: Soticlestat; Test type: Superiority; p = 0.540, t-test, 2 sided — The p-values were estimated using a two-sample t-test

8. Secondary Outcome: Percent Change From Baseline in CSS at the End of Part A
Description: Signs and symptoms reflecting the sensory, vasomotor, sudomotor/edema, and motor/trophic disturbances of CRPS had been incorporated into a clinically feasible CSS. Total CSS is a 16-point score which was calculated by the number of "yes" answers to the questions on the 8 symptoms and 8 signs when all 16 questions were answered. Negative percent change from Baseline indicates improvement.
Time Frame: Baseline and Week 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Double-Blind Treatment Period - Part A: Placebo | Double-Blind Treatment Period - Part A: Soticlestat
Number analyzed (Participants) | 6 | 13
percent change | -16.1 (18.89) | -23.8 (26.29)

ADVERSE EVENTS:
Time Frame: From signing of the informed consent up to 15 days after last dose of the study drug (Up to approximately Week 32)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Double-Blind Treatment Period - Part A: Placebo | Double-Blind Treatment Period - Part A: Soticlestat | Open-Label Extension Period - Part B: Soticlestat
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/15 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/9 | 3/15 | 0/18
Other Adverse Events (participants affected / at risk) | 9/9 | 12/15 | 10/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Treatment Period - Part A: Placebo (N=9) | Double-Blind Treatment Period - Part A: Soticlestat (N=15) | Open-Label Extension Period - Part B: Soticlestat (N=18)
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Treatment Period - Part A: Placebo (N=9) | Double-Blind Treatment Period - Part A: Soticlestat (N=15) | Open-Label Extension Period - Part B: Soticlestat (N=18)
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 2 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 1
Fatigue (General disorders) | 0 | 2 | 0
Influenza like illness (General disorders) | 0 | 2 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 4 | 0
Headache (Nervous system disorders) | 4 | 2 | 5
Lethargy (Nervous system disorders) | 1 | 1 | 0
Depressed mood (Psychiatric disorders) | 2 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 2 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Study Protocol (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT03990649/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/49/NCT03990649/SAP_001.pdf